CLINICAL TRIAL: NCT00485680
Title: Olanzapine Versus Lithium Carbonate in the Treatment of Bipolar Disorder, Manic or Mixed Episodes
Brief Title: Olanzapine Versus Comparator in the Treatment of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7598; F1D-GH-LOBV
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — olanzapine-fluoxetine combination; Lithium Carbonate

INTERVENTIONS:
Drug: Olanzapine Hydrochloride
Drug: Lithium Carbonate

SUMMARY:
The purpose of this trial is compare the efficacy of olanzapine and Lithium Carbonate in the treatment of bipolar disorder, manic or mixed episodes, in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in- or out-patients at least 18 years of age
* Patient must have a diagnosis of bipolar I disorder and currently display acute manic or mixed episodes (with or without psychotic features) according to the DSM-IV based on clinical assessment
* Patients must have a level of understanding sufficient to agree to all tests and examinations required by the protocol
* Patients must have a Y-MRS total score of greater than or equal to 20 at both visits 1 & 2
* Patients must be considered reliable

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months
* Current or past diagnosis of schizophrenia or other psychotic disorder (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV
* Documented history of intolerance to olanzapine or Lithium Carbonate
* Treatment with clozapine within 4 weeks prior to visit 2. Treatment with other antipsychotic drugs or mood stabilizers within 2 days prior to visit 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-12; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Investigate the efficacy of olanzapine once a day orally for 4 weeks to Lithium Carbonate orally in the treatment of Chinese patients with bipolar I disorder, manic or mixed episodes, with or without psychotic features as measured by the CGI-BP Severity

SECONDARY OUTCOMES:
Assess the efficacy of olanzapine compared with Lithium Carbonate in improving clinical symptomatology in patients diagnosed with bipolar disorder, manic or mixed episodes after acute treatment as measured by the Y-MRS
Assess the efficacy of olanzapine compared with Lithium Carbonate in improving clinical symptomatology in patients diagnosed with bipolar disorder, manic or mixed episodes after acute treatment as measured by the BRPs, MADRS.
Assess the safety of olanzapine compared with Lithium Carbonate. Treatment-emergent adverse events, change in vital signs, laboratory analytes and ECG will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai, China

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com